CLINICAL TRIAL: NCT01464723
Title: VEGF and HTRA1 DNA Polymorphisms in Neovascular AMD Pathogenesis and Response to Lucentis
Brief Title: Study EvAluating Genotypes While Using Lucentis 2
Acronym: SEAGUL2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080693
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lucentis (Experimental): Consented, enrolled subjects will receive multiple open-label intravitreally administered 0.5 mg ranibizumab administered monthly for the first 4 months, and then as needed for a total duration of 12 months.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injections of 0.5 mg ranibizumab administered monthly for the first 4 months, and then as needed for a total duration of 12 months.
  Other Names: Lucentis

SUMMARY:
The purpose of the study is to investigate whether the efficacy of Lucentis treatment for exudative age-related macular degeneration is associated with VEGF and HTRA1 DNA polymorphisms

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a progressive disease that causes irreversible visual impairment and blindness in nearly 50 million people globally. Although geographic atrophy and neovascularization represent the advanced forms of AMD, neovascular AMD is the more aggressive form and accounts for almost 90% of blindness from this disease. It is characterized by choroidal neovascularization (CNV) which is the development of abnormal blood vessels underneath the retina. Randomized clinical trials (MARINA, ANCHOR) have conclusively demonstrated that continued intravitreal therapy with Lucentis (ranibizumab) in patients with subfoveal CNV from AMD leads to stabilization of vision in over 90% of patients and improvement in vision in at least a third of the patients and has led to the approval of Lucentis for the treatment of neovascular AMD (see investigator brochure). This study could provide insight as to the reasons that some patients do not experience vision stabilization with Lucentis, and could possibly help physicians to determine which patients are the best candidates for receiving Lucentis.

This is an open-label study of 100 treatment-naïve (study eye only) AMD patients treated on-label with intravitreally administered Lucentis. Consented, enrolled subjects will receive multiple open-label intravitreal injections of 0.5 mg ranibizumab administered monthly for the first 4 months, and then as needed for a total duration of 12 months. Their blood will be genotyped and sequenced for various SNPs on VEGF and HTRA1.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with the study assessments for the full duration of the study.
* Age > 50 years.
* Treatment naïve (study eye only) AMD patients that are determined to be candidates for ranbizumab.
* Visual acuity 20/32 to 20/230.

Exclusion Criteria:

* Pregnancy
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Previous therapy in study eye for AMD or other retinal disease which may be used in the treatment of AMD.
* Any other condition that the investigator believes would pose a significant hazard to the subject if on-label ranibizumab were prescribed
* Any participation in another simultaneous medical investigation or trial for AMD *Concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy, advanced glaucoma)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shiley Eye Center, University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Data not available for sharing.

REFERENCES:
- [Derived] Zhao L, Grob S, Avery R, Kimura A, Pieramici D, Lee J, Rabena M, Ortiz S, Quach J, Cao G, Luo H, Zhang M, Pei M, Song Y, Tornambe P, Goldbaum M, Ferreyra H, Kozak I, Zhang K. Common variant in VEGFA and response to anti-VEGF therapy for neovascular age-related macular degeneration. Curr Mol Med. 2013 Jul;13(6):929-34. doi: 10.2174/15665240113139990048. PMID 23745581

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Principal Investigator has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful due to all study team members having left the University. No study data are available, attempts were made to find the data but were unsuccessful.
Groups:
- Lucentis: Consented, enrolled subjects will receive multiple open-label intravitreally administered 0.5 mg ranibizumab administered monthly for the first 4 months, and then as needed for a total duration of 12 months.
  Ranibizumab : Intravitreal injections of 0.5 mg ranibizumab administered monthly for the first 4 months, and then as needed for a total duration of 12 months.
Period: Overall Study
Arm/Group | Lucentis
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Principal Investigator has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful due to all study team members having left the University. No study data are available, attempts were made to find the data but were unsuccessful.
Arm/Group | Lucentis
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Genotype at VEGF and HTRA1 SNPs of Patients Gaining ≥ 0 Letters of Visual Acuity in Response to Ranibizumab Treatment Over a 4 Month Period.
Time Frame: 5 years
Population: as for baseline characteristics
Arm/Group | Lucentis
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Genotype at VEGF and HTRA1 SNPs of Patients Who Lose Visual Acuity (Gain <0 Letters) at 4, 6 and 12 Months After Initial Treatment.
Time Frame: 5 years
Population: as for baseline characteristics
Arm/Group | Lucentis
Number analyzed (Participants) | 0

3. Secondary Outcome: To Determine Whether Change in Retinal Thickness is Correlated With Genotype
Time Frame: 5 years
Population: as for baseline characteristics
Arm/Group | Lucentis
Number analyzed (Participants) | 0

4. Secondary Outcome: To Determine the Mean Number of Injections Per Year Patients in the Study Require.
Time Frame: 5 years
Population: as for baseline characteristics
Arm/Group | Lucentis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The Principal Investigator has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful due to all study team members having left the University. No study data are available, attempts were made to find the data but were unsuccessful.
Arm/Group | Lucentis
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful due to all study team members having left. No study data are available, attempts were made to find the data but were unsuccessful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No